CLINICAL TRIAL: NCT00357435
Title: Clinical and Molecular Studies in Families With Corneal Dystrophy or Other Inherited Corneal Diseases
Brief Title: Studies in Families With Corneal Dystrophy or Other Inherited Corneal Diseases
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040008; 04-EI-0008
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2016-07-21

CONDITIONS: Corneal Dystrophies, Hereditary; Corneal Disease
Keywords: Cornea; Genetics; Dystrophy; Gene; Mapping; Molecular; Bietti; Fleck; Positional Cloning; Linkage
MeSH Terms: conditions — Corneal Dystrophies, Hereditary; Corneal Diseases

SUMMARY:
This study will explore the clinical and hereditary (genetic) features of corneal dystrophy and other inherited corneal disease. Corneal dystrophy is clouding of the cornea - the transparent part of the eye covering the iris and pupil that passes light to the back of the eye. When the cornea becomes cloudy, interfering with the passage of light, vision may be impaired or lost. Corneal problems may occur with vision problems alone, or with other problems, such as changes in facial appearance or bone or joint problems. A better understanding of these genetic conditions may help in the development of better diagnostic tests and methods of disease management.

Patients with corneal dystrophies and related corneal disease and their family members may be eligible for this study. Participants will be drawn from patients enrolled in other studies of corneal dystrophy at the NEI and collaborating clinics.

Participants will undergo the following tests and procedures:

* Medical and surgical history
* Verification of diagnosis
* Construction of a family tree regarding familial vision problems
* Complete eye examination, including dilation of the pupils and photography of the cornea, tests of color vision, field of vision, and the ability to see in the dark, and photographs of the eye.
* Blood sample collection to identify the genes responsible for corneal disease and ascertain how they cause disease.

DETAILED DESCRIPTION:
Objective: This project, Clinical and Molecular Studies in Families With Corneal Dystrophy or Other Inherited Corneal Diseases will study the inheritance of corneal dystrophy and other inherited corneal diseases, both Mendelian and complex in order to identify the genes that, when mutated, cause corneal disease and the pathophysiology through which they act.

Study Population: Families of many nationalities and ethnic backgrounds. We will study a maximum or 2,000 patients and family members.

Design: The study consists of ascertaining individuals, and especially families with multiple individuals, affected by corneal dystrophy and other inherited corneal diseases. These patients and their families will undergo detailed ophthalmological examinations to characterize their corneal disease and determine their affectation status. A blood sample will be collected from each individual for isolation of DNA and in some individuals for lymphoblastoid transformation to establish a renewable source of DNA. Linkage analysis, physical mapping, and mutational screening will be carried out to identify the specific the gene and the mutations in it that are associated with corneal disease in this family. If necessary, the gene product will be characterized biochemically. All associate investigators will carry out patient ascertainment, diagnosis, and sample referral, and in some cases molecular genetic analyses. The study will enroll subjects at NEI and collaborating institutions.

Outcome Measures: Linkage will be determined using the lod score method and mutations in specific genes will be assessed using a combination of residue conservation, blosum score, and molecular modeling. Biochemical, metabolic, and physiological effects will be individualized to the specific assay.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects with the following will be recruited:

1. Individuals or family members of individuals with corneal dystrophies and related corneal diseases.
2. Adults must be capable of providing their own consent.
3. All subjects must be able to cooperate with study examination and phlebotomy.
4. Older than 4 years of age.

EXCLUSION CRITERIA:

1. Diseases, infections, or trauma that mimic corneal diseases.
2. Children requiring sedation for study procedures.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2003-10-06; Study Completion 2016-07-21

CONTACTS AND LOCATIONS:
Overall Officials: James F Hejtmancik, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (6):
- United States (4):
  - Jules Stein Eye Institute, UCLA, Los Angeles, California
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas, Houston, Houston, Texas
- Zhongshan Opthalmic Center, Guangzhou, China
- Seconda Universita degli, Naples, Italy

REFERENCES:
- [Background] Klintworth GK, Sommer JR, Obrian G, Han L, Ahmed MN, Qumsiyeh MB, Lin PY, Basti S, Reddy MK, Kanai A, Hotta Y, Sugar J, Kumaramanickavel G, Munier F, Schorderet DF, El Matri L, Iwata F, Kaiser-Kupfer M, Nagata M, Nakayasu K, Hejtmancik JF, Teng CT. Familial subepithelial corneal amyloidosis (gelatinous drop-like corneal dystrophy): exclusion of linkage to lactoferrin gene. Mol Vis. 1998 Dec 31;4:31. PMID 9873069
- [Background] Lee J, Jiao X, Hejtmancik JF, Kaiser-Kupfer M, Chader GJ. Identification, isolation, and characterization of a 32-kDa fatty acid-binding protein missing from lymphocytes in humans with Bietti crystalline dystrophy (BCD). Mol Genet Metab. 1998 Oct;65(2):143-54. doi: 10.1006/mgme.1998.2723. PMID 9787106
- [Background] Jiao X, Munier FL, Iwata F, Hayakawa M, Kanai A, Lee J, Schorderet DF, Chen MS, Kaiser-Kupfer M, Hejtmancik JF. Genetic linkage of Bietti crystallin corneoretinal dystrophy to chromosome 4q35. Am J Hum Genet. 2000 Nov;67(5):1309-13. doi: 10.1016/S0002-9297(07)62960-7. Epub 2000 Sep 21. PMID 11001583